CLINICAL TRIAL: NCT00593931
Title: Development Of New Techniques For Functional Magnetic Resonance Imaging Of The Brain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator is deceased
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200210591
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Diagnosis, Psychiatric
Keywords: Brain functional MRI
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Normal Subjects
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — Functional Magnetic Resonance Imaging without contrast

SUMMARY:
This Protocol is intended to facilitate development and testing of new techniques for functional MRI by UC Davis Research Faculty, as well as to facilitate the evaluation of new techniques provided by the system manufacturers (GE and Siemens).

DETAILED DESCRIPTION:
New techniques covering a wide range of clinical and scientific applications will be developed, tested and evaluated. These include 1. Investigation of sensory stimulus processing and cognitive processing, both in normal subjects and patients with psychiatric disorders, 2. Early detection of stroke and other ischemic injury, and 3. Characterization of tumor distribution and activity. The new techniques will routinely need to be tested with respect to the following: 1. Sensitivity to blood oxygenation versus blood flow versus blood volume contrast mechanisms, 2. Signal-to-noise and contrast-to-noise ratio, 3. Spatial and temporal resolution, 4. Distribution and severity of image artifacts, and 5. Duty cycle limitations. Most clinical applications will require coverage of the entire brain and consequently high duty cycle operation, which needs to be traded off with spatial and temporal resolution, as well as contrast mechanisms. The work will also involve the testing of different experimental paradigms (time sequence of stimuli or cognitive tasks) to identify that which provides the highest signal change associated with the specific brain activity of interest.

Although 3T provides twice the signal of 1.5T systems, for some research applications this image quality advantage of 3T may be outweighed by other effects of higher field on the signal. Consequently, most new techniques will be evaluated on both the 1.5T and 3T systems, and a decision will be made based upon the overall image quality, regarding which system is to be used.

The Protocol does not involve injection of any contrast agent or drug, or other minimally-invasive or invasive procedure. It is intended specifically for those studies in which the subject is required, in addition to trying to relax and lie still, only to experience and respond to various non-harmful sensory stimuli, or to perform common cognitive (e.g. math calculations) and or motor (e.g. finger tapping) tasks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* ability to give informed, written consent
* Not pregnant or breastfeeding

Exclusion Criteria:

* Electrically, magnetically, or mechanically activated implants (for example, cardiac-pacemakers)
* Ferromagnetic implant, such as an aneurysm clip, surgical clip, or prosthesis
* History of uncontrolled claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 1999-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
transient changes in blood flow in the brain that occurs with neuronal activity | Post-scanning

SECONDARY OUTCOMES:
Sensitivity to blood oxygenation versus blood flow versus blood volume contrast mechanisms | Post-scanning

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Buonocore, M.D., Ph.D., Principal Investigator — UC Davis Dept. of Radiology